CLINICAL TRIAL: NCT06419699
Title: Responsiveness and the Minimal Clinically Important Difference of the Chelsea Critical Care Physical Assessment Tool (CPAx) in Critically Ill, Mechanically Ventilated Adults
Brief Title: CPAx: Responsiveness and Minimal Clinically Important Difference
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 5678
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Muscle Weakness; Critical Illness Myopathy; Critical Illness Polyneuropathy; Critical Illness Polyneuromyopathy; Physical Inactivity
Keywords: Physiotherapy; Physical function and activity; Early rehabilitation; Measurement instrument; Critical illness; Critical care outcomes
MeSH Terms: conditions — Muscle Weakness; Polyneuropathies; Sedentary Behavior; Motor Activity; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive care unit (ICU) acquired weakness is a common complication associated with long-term physical impairments in survivors of a critical illness. The Chelsea Critical Care Physical Assessment tool (CPAx) is a valid and reliable instrument for physical function and activity in critically ill patients at risk for muscle weakness. However, its ability to measure change over time (responsiveness) and the minimal clinically important difference (MCID) have not yet been rigorously investigated. This multi-centre, mixed-methods, longitudinal cohort study therefore aims to establish responsiveness and the MCID of the CPAx in the target population from ICU baseline to ICU and hospital discharge. The study uses routine data from standard physiotherapy sessions like mobility, function and activity with no additional burden for critically ill adults. The investigators expect the CPAx to be responsive allowing its use as a primary outcome in future effectiveness trials for the treatment of ICU-acquired weakness using the newly established MCID for sample size calculation. A high quality, rigorously tested measurement tool for physical function and activity in the ICU should benefit researchers, clinicians and patients.

DETAILED DESCRIPTION:
The use of invasive life support in critically ill patients clearly saves lives but carries substantial risks, including intensive care unit (ICU) acquired weakness and long-term disability. The investigators urgently need a valid, reliable, and responsive measurement tool for this population to use in clinical practice and trials. The Chelsea Critical Care Physical Assessment tool (CPAx) is a promising measurement instrument to measure change in critically ill patients' physical function and activity. After several studies have confirmed its validity and excellent reliability, it is time to confirm responsiveness and to establish the MCID in a large, international sample of the target population. This multi-centre, mixed-methods, longitudinal cohort study will include critically ill, mechanically ventilated (>72h) adults at risk for muscle weakness and collect their mobility, physical function and activity with the CPAx and other relevant measures at ICU baseline, to ICU and hospital discharge. Responsiveness will be determined by the ability of the CPAx to identify change according to a prespecified anchor (criterion validity) and by testing prospective hypotheses about the expected magnitude of change between the CPAx and other relevant measures (construct validity). The MCID will be established with anchor- and distribution-based methods, whereby a seven-point global rating of change scale obtained from treating ICU physiotherapists will serve as anchor to distinguish improved from unchanged patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mechanical ventilation ≥ 72 hours
* Expected to remain for ≥ 48 hours in the ICU
* Physiotherapy referral

Exclusion Criteria:

* Not expected to survive to hospital discharge (imminent to death)
* Second or subsequent ICU admission for this hospital stay
* Transfer from external ICU (with an ICU stay of >72 hours)
* Primary neurological admission diagnosis (i.e., of the central nervous system including stroke, intracerebral haemorrhage, traumatic brain injury)
* Known pregnancy
* Living in a care facility pre-admission (severe pre-existing mental or physical disability)
* Local regulations (i.e. Switzerland: refusal of general consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population are critically ill adults who are mechanically ventilated for a prolonged period (≥ 72 hours) and who have an increased risk for ICUAW and long-term impairment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Chelsea Critical Care Physical Assessment tool (CPAx) change score | Assessed at ICU discharge (within 24 hours before or after ICU discharge)
  CPAx change score for ICU period (ICU baseline to ICU discharge); CPAx ranges from 0 (worst score) to 50 (best score)

SECONDARY OUTCOMES:
CPAx change score | Assessed at hospital discharge (last value before discharge)
  CPAx change score for hospital period (ICU to hospital discharge); CPAx ranges from 0 (worst score) to 50 (best score)
Global rating of change scale | ICU and hospital discharge (change for ICU and hospital period)
  Seven-point global rating of change scale (GRC): (1) very much improved; (2) much improved; (3) little improved; (4) no change; (5) little deterioration; (6) much deterioration; (7) very much deterioration for 'physical function and activity' (rated by treating physiotherapist)
ICU Mobility Scale | ICU baseline (within 72-144h after ICU admission), ICU and hospital discharge
  To evaluate mobility level, the score ranges from 0 (worst) to 10 (best)
Medical Research Council Sum Score | ICU baseline (within 72-144h after ICU admission), ICU and hospital discharge
  To assess muscle strength, the minimal score is 0 (worst), the maximal score 60 (best), ICUAW is defined as <48 points
Richmond Agitation-Sedation Scale | ICU baseline (within 72-144h after ICU admission), ICU and hospital discharge
  To assess the level of sedation and/or cooperation, score ranges from -5 (unarousable) to +4 (combative)
Modified Iowa Level of Assistance Scale | ICU baseline (within 72-144h after ICU admission), ICU and hospital discharge
  To determine assistance in functional tasks, the score ranges from 0 (worst) to 36 (best)
ICU and discharge destinations | ICU and hospital discharge
  Categorical variable (death, external/internal hospital ward, external ICU/hospital, rehabilitation, home, other) to assess the predictive validity of the CPAx score

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Eggmann, PhD, Principal Investigator — Inselspital, Bern University Hospital, Switzerland; Monash University, Australia
Locations (3):
- Australia (2):
  - Monash Health, Clayton
  - Alfred Health, Melbourne
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Solely anonymised main outcome data

REFERENCES:
- [Background] Corner EJ, Wood H, Englebretsen C, Thomas A, Grant RL, Nikoletou D, Soni N. The Chelsea critical care physical assessment tool (CPAx): validation of an innovative new tool to measure physical morbidity in the general adult critical care population; an observational proof-of-concept pilot study. Physiotherapy. 2013 Mar;99(1):33-41. doi: 10.1016/j.physio.2012.01.003. Epub 2012 Mar 30. PMID 23219649
- [Background] Eggmann S, Verra ML, Stefanicki V, Kindler A, Seyler D, Hilfiker R, Schefold JC, Bastiaenen CHG, Zante B. German version of the Chelsea Critical Care Physical Assessment Tool (CPAx-GE): translation, cross-cultural adaptation, validity, and reliability. Disabil Rehabil. 2022 Aug;44(16):4509-4518. doi: 10.1080/09638288.2021.1909152. Epub 2021 Apr 19. PMID 33874842
- [Background] Eggmann S, Verra ML, Stefanicki V, Kindler A, Schefold JC, Zante B, Bastiaenen CHG. Predictive validity of the Chelsea Critical Care Physical Assessment tool (CPAx) in critically ill, mechanically ventilated adults: a prospective clinimetric study. Disabil Rehabil. 2023 Jan;45(1):111-116. doi: 10.1080/09638288.2021.2022785. Epub 2022 Jan 7. PMID 34994664
- [Derived] Eggmann S, Paton M, Villinger C, Bradley S, Hellings T, Hills A, Venetz P, Broadley T, Charles-Nelson A, Hodgson C. Responsiveness and the minimal clinically important difference of the Chelsea Critical Care Physical Assessment tool (CPAx) in critically ill, mechanically ventilated adults: a study protocol for a prospective, multicentre, cohort study. BMJ Open. 2025 Sep 18;15(9):e102374. doi: 10.1136/bmjopen-2025-102374. PMID 40973373